CLINICAL TRIAL: NCT02877017
Title: Family Activation and Communication About Errors and Safety (FACES)
Acronym: FACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alisa Khan, Assistant Professor, Pediatrics, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-P00022336
Record Dates: First submitted 2016-08-17; First posted 2016-08-24 (Estimated); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Family Reported Errors and Adverse Events

STUDY DESIGN:
Intervention Model Description: pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention arm (No Intervention): This arm is the pre-intervention arm of parents and providers before the family safety reporting bundle has been implemented.
- Post-intervention arm (Experimental): This arm is the post-intervention arm of parents and providers after the family safety reporting bundle has been implemented on the study units.
  Interventions: Behavioral: Family safety reporting intervention

INTERVENTIONS:
Behavioral: Family safety reporting intervention — family safety reporting intervention for families and providers
  Arms: Post-intervention arm

SUMMARY:
Miscommunications are a leading cause of serious medical errors in hospitals, contributing to more than 60% of sentinel events, the most serious adverse events reported to the Joint Commission. Efforts to improve patient safety in hospitals have centered on improving communication between providers. While provider-focused communication interventions have led to reductions in patient harm, patients and families have been notably absent from most interventions to improve patient safety. This proposal seeks to develop a family safety reporting intervention.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of a child hospitalized on the study units during the study period or hospital employee who works on the study unit(s)
* Country of Origin: United States
* Primarily English- or Spanish-speaking

Exclusion Criteria:

* International patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 985 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alisa Khan, MD, MPH, Principal Investigator — Boston Children's Hospital/Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol enrollment reflects participants who are families of hospitalized children and providers among the hospital units. The Participant Flow reflects only families of hospitalized children that participated in the mobile tool aspect of the intervention, which the "Providers" group did not participate in and therefore are not included here.
Groups:
- Pre-intervention Arm: This arm is the pre-intervention arm of participants before the family safety reporting bundle has been implemented.
- Post-intervention Arm: This arm is the post-intervention arm of participants after the family safety reporting bundle has been implemented on the study units.
  Family safety reporting intervention: family safety reporting intervention for families and providers
Period: Overall Study
Arm/Group | Pre-intervention Arm | Post-intervention Arm
Started | 232 | 208
Completed | 207 | 157
Not Completed | 25 | 51

BASELINE CHARACTERISTICS:
Population: English- and Spanish-speaking parents of hospitalized children with medical complexity (CMC). Baseline data for providers and hospitalized children was not collected because the intervention was being conducted with the families of hospitalized children, and not providers or hospitalized children. Missing data from participants may occur as some participants did not provide all baseline information.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-intervention Arm | Post-intervention Arm | Total
Number analyzed (Participants) | 207 | 157 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We enrolled 440 participants overall (pre-intervention=232, post-intervention=208). Of these, 364 (82.7%) completed surveys (pre-intervention=207, post-intervention=157).
  years | 48 (11) | 45 (10) | 46 (11)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We enrolled 440 participants overall (pre-intervention=232, post-intervention=208). Of these, 364 (82.7%) completed surveys (pre-intervention=207, post-intervention=157).
  Participants
    number analyzed (Participants) | 205 | 155 | 360
    Female | 168 | 134 | 302
    Male | 37 | 21 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: We enrolled 440 participants overall (pre-intervention=232, post-intervention=208). Of these, 364 (82.7%) completed surveys (pre-intervention=207, post-intervention=157).
  Participants
    number analyzed (Participants) | 205 | 155 | 360
    American Indian or Alaskan Native, Non- Hispanic | 1 | 0 | 1
    Asian/Pacific Islander, non-Hispanic | 5 | 4 | 9
    Black/African-American, non-Hispanic | 9 | 9 | 18
    Hispanic | 30 | 34 | 64
    Multi-racial, non-Hispanic | 4 | 1 | 5
    Other, non-Hispanic | 4 | 2 | 6
    White, non-Hispanic | 152 | 105 | 257
Region of Enrollment [Count of Participants; unit: Participants] — Population: We enrolled 440 participants overall (pre-intervention=232, post-intervention=208). Of these, 364 (82.7%) completed surveys (pre-intervention=207, post-intervention=157).
  Participants
    United States | 207 | 157 | 364
English Proficiency [Count of Participants; unit: Participants] — Population: We enrolled 440 participants overall (pre-intervention=232, post-intervention=208). Of these, 364 (82.7%) completed surveys (pre-intervention=207, post-intervention=157).
  Participants
    number analyzed (Participants) | 205 | 154 | 359
    Proficient | 174 | 132 | 306
    Limited English Proficient | 31 | 22 | 53
Education Attainment [Count of Participants; unit: Participants] — Population: We enrolled 440 participants overall (pre-intervention=232, post-intervention=208). Of these, 364 (82.7%) completed surveys (pre-intervention=207, post-intervention=157).
  Participants
    number analyzed (Participants) | 206 | 155 | 361
    Less than college | 105 | 85 | 190
    Completed college or higher | 101 | 70 | 171

OUTCOME MEASURES:

1. Primary Outcome: Family Safety Reporting Rates
Description: Our primary outcome was family-reported safety concerns, defined as reporting safety concern(s) via pre-discharge survey (baseline and intervention) or mobile tool (intervention). Safety concerns were counted once if reported both via survey and mobile tool.
Time Frame: During both baseline and intervention periods, the time frame for each participant being assessed was from admission to discharge, on average approximately 5-14 days.
Population: We included English/Spanish-speaking parents of patients of all ages hospitalized on the complex care service.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-intervention Arm | Post-intervention Arm
Number analyzed (Participants) | 207 | 157
Participants | 61 | 60

2. Secondary Outcome: Family Reported Hospital Safety Climate Scores
Description: For Family Reported Hospital Safety Climate Scores, Child HCAHPS safety experience was used to ask whether hospital staff told participants how to report concerns about mistakes. We examined top-box (top-most, e.g., 5 of 5, Likert scale) safety climate scores baseline vs intervention and proportion of parents reporting "yes definitely" or "yes somewhat" vs "no" to the Child HCAHPS "tell you how to report" question.
Time Frame: as for outcome 1
Population: We included English/Spanish-speaking parents of patients of all ages hospitalized on the complex care service.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-intervention Arm | Post-intervention Arm
Number analyzed (Participants) | 182 | 151
Participants | 66 | 69

ADVERSE EVENTS:
Time Frame: Time on study unit, from admission to discharge, on average approximately 9 days.
Description: Documented system-wide adverse event reports were reviewed and evaluated on a weekly basis. Of note, we collected adverse events as part of this study's primary outcome and all the events reported below are unrelated to the study intervention. We collected events through family safety reporting and hospital collected events which were then chart reviewed.
Groups:
- Pre-intervention Arm: This arm is the pre-intervention arm of participants (families of children with medical complexity) whose children had monitored/assessed adverse events before the family safety reporting bundle had been implemented on the study units.
- Post-intervention Arm: This arm is the post-intervention arm of participants (families of children with medical complexity) whose children had recorded adverse events after the family safety reporting bundle had been implemented on the study units.
Arm/Group | Pre-intervention Arm | Post-intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/232 | 0/208
Serious Adverse Events (participants affected / at risk) | 0/232 | 0/208
Other Adverse Events (participants affected / at risk) | 14/232 | 23/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-intervention Arm (N=232) | Post-intervention Arm (N=208)
Serious Adverse Events (General disorders) | 0 (0) | 0 (0) — Serious Adverse Events were those that we rated categories G and H using the NCC MERP Index.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-intervention Arm (N=232) | Post-intervention Arm (N=208)
Other Adverse Events (Cardiac disorders) | 1 | 0 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Gastrointestinal disorders) | 2 | 2 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Infections and infestations) | 2 | 2 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Injury, poisoning and procedural complications) | 2 | 5 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Musculoskeletal and connective tissue disorders) | 0 | 1 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Nervous system disorders) | 3 | 10 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Product Issues) | 0 | 1 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Renal and urinary disorders) | 1 | 0 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Skin and subcutaneous tissue disorders) | 2 | 0 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.
Other Adverse Events (Surgical and medical procedures) | 1 | 2 — Other Adverse Events were those that we rated categories E and F using the NCC MERP Index.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT02877017/Prot_SAP_000.pdf